CLINICAL TRIAL: NCT00752011
Title: Phase I Dose Escalating Study Of Tas-106 In Combination With Carboplatin In Patients With Solid Tumors
Brief Title: Phase I Study of TAS-106 in Combo With Carboplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0623
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Cancer; Solid Tumors
Keywords: Cancer; Solid Tumors; Advanced Cancer; Carboplatin; Paraplatin; TAS-106; Antitumor Activity; Biomarkers
MeSH Terms: conditions — Neoplasms | interventions — 1-(3-C-ethynylribopentofuranosyl)cytosine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin + TAS-106 (Experimental): Carboplatin starting dose AUC of 4, administered by vein over 60 minutes, Day 1 of 3 Week Cycle. TAS-106 starting dose 2.0 mg/m^2 by vein over 24 hours, Day 1 of 3 Week Cycle.
  Interventions: Drug: TAS-106; Drug: Carboplatin

INTERVENTIONS:
Drug: TAS-106 — Starting dose 2.0 mg/m^2 by vein over 24 hours, Day 1 of 3 Week Cycle.
Drug: Carboplatin — Starting dose AUC of 4, administered by vein over 60 minutes, Day 1 of 3 Week Cycle.
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the combination of TAS-106 and carboplatin that can be given to patients with advanced cancer or cancer that has spread.

Objectives:

Primary Objectives:

To determine the maximum tolerated dose (MTD) of the combination of TAS-106 and carboplatin administered by intravenous infusion every 3 weeks.

To perform Pharmacokinetic (PK) analysis of TAS-106 and carboplatin

Secondary objectives:

To assess the antitumor activity of TAS-106 combined with carboplatin

To investigate the relationship between selected biomarkers and efficacy and safety outcomes.

DETAILED DESCRIPTION:
The Study Drugs:

TAS-106 and carboplatin are designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the study drug combination that is based on when you joined this study. Up to 6 dose levels of the study drug combination will be tested. Three (3) participants will be enrolled at each dose level. If no intolerable side effects occur in the first group of 3 people, the next 3 people enrolled in the study will receive the same dose of carboplatin and a higher dose of TAS-106. If this second group has no intolerable side effects, the next 3 people will receive a higher dose of carboplatin while receiving the same dose of TAS-106 as the second group. This will continue until the highest safe dose combination is found.

Study Drug Administration:

A "cycle" in this study is 3 weeks long. On Day 1 of each cycle, you will receive carboplatin by vein over 60 minutes, followed by TAS-106 by vein over 24 hours.

Study Visits:

On Day 1 of each cycle (+/- 1 day), you will come to the clinic to have the following procedures performed:

* You will have a complete physical exam, including measurement of vital signs and weight.
* You will have a neurological exam.
* You will be asked about any drugs you have taken recently and any side effects you may have experienced. The study doctor may give you drugs to lessen any possible side effects.
* You will have a performance status evaluation.
* Blood (about 3 teaspoons) and urine will be collected for routine tests.

On Day 1 of Weeks 2 and 3 of each cycle (+/- 3 days), blood (about 3 teaspoons) will be drawn for routine tests. If your blood cell counts (white blood cells, red blood cells, and/or platelets) drop to a low level, you may need to have these routine tests repeated more often than once a week.

At the end of every 2 cycles (+/- 1 week), you will have CT scans, MRI scans, and/or x-rays to check the status of the disease.

You must stay in the Houston area during Cycle 1. During that time, all blood tests and other study tests and procedures must be done at MD Anderson. Starting in Cycle 2, if you prefer, you may have the blood tests at Weeks 2 and 3 of each cycle performed at a medical laboratory that is close to your home. If you need to have the additional blood cell count testing performed as well, those blood tests can also be done close to home. All other study tests and procedures must be done at M. D. Anderson.

Length of Study Participation:

You may continue to stay on the study drugs for as long as you are benefiting. If the cancer gets worse or you experience intolerable side effects, you will be taken off study. If you experience side effects that are severe but not intolerable, however, your doctor may decide that it is necessary to delay your next dose of the study drug combination and/or lower the dose.

End-of-Study Visit:

When you go off study for any reason, you will have an end-of-study visit with all of the same tests performed as at your other study visits. You will also have an ECG.

This is an investigational study. Carboplatin is FDA approved and commercially available for other uses. TAS-106 is not FDA approved or commercially available. The combination of carboplatin and TAS-106 is not FDA approved or commercially available. At this time, the combination is being used in research only.

Up to 55 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of a solid tumor. Advanced or metastatic disease that is refractory to standard therapy or for which no standard therapy exists
2. Objective evidence or disease recurrence or metastatic disease
3. Age >/= 18 years old at study entry
4. Measurable or evaluable disease
5. A score of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
6. Hemoglobin > 9.0 g/dL; Platelet count >/=100,000/uL; Absolute neutrophil count (ANC) >/=1500/uL
7. Serum creatinine </=1.5 mg/dL; if > 1.5mg/dL, then a calculated creatinine clearance must be >/=60 mL/min
8. Total bilirubin </=1.5 mg/dl; ALT </= 2 times the upper limit of normal (ULN) (may be </= 5 times ULN if due to metastatic disease in the liver).
9. Fertile men and women, and their partners, must use a medically effective contraception method (spermicide with male or female condoms, cervical sponge, IUD, cervical cap, or diaphragm or oral, implantable, transdermal, or injectable contraceptives) throughout the treatment period and for 30 days after the last dose of study medication. Premenopausal women of reproductive capacity and women less than 12 months after menopause must have a negative pregnancy test documented prior to study entry.
10. Signed written informed consent per institutional and federal regulatory requirements.

Exclusion Criteria:

1. Has known hypersensitivity to carboplatin
2. Radiological or clinical evidence of brain involvement or leptomeningeal disease
3. Have history of Human Immunodeficiency Virus, hepatitis B, or hepatitis C infection
4. >/=grade 2 peripheral neuropathy
5. Women who are pregnant or breast feeding.
6. Serious illness or medical condition(s) including but not limited to the following: a) Congestive heart failure or uncontrolled angina pectoris. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or dysrhythmias. b) Active infection. c) Unstable diabetes mellitus. d) Psychiatric disorder that may interfere with consent and/or protocol compliance
7. Female or male subject of reproductive capacity who is unwilling to use methods appropriate to prevent pregnancy during the course of this study.
8. Receiving concurrent chemotherapy, investigational agents radiotherapy, or surgery.
9. Received radiation therapy to >30% of bone marrow (e.g., whole of pelvis or half of spine).
10. Received any investigational drug within the last 30 days.
11. Not fully recovered from any prior surgery (at least 4 weeks recovery period for major surgery), and from any reversible side effects related to the administration of cytotoxic chemotherapy, investigational agents, or radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-06; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | With every 3 week cycle

SECONDARY OUTCOMES:
To review relationship between selected biomarkers and efficacy/safety outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: U.T. M.D. Anderson Cancer Center website — http://www.mdanderson.org